CLINICAL TRIAL: NCT07314541
Title: A Phase Ia, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Tolerability of KMY Tablets in Healthy Subjects
Brief Title: A Phase Ia Study of KMY Tablets in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lei Yunshang Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2025-CP-KMY-01
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KMY Tablets (Experimental): Participants will receive the active drug, KMY tablet. The study consists of three parts:
  Part A (Single Ascending Dose): Participants will be assigned to one of eight predefined dose cohorts (2, 6, 10, 20, 40, 60, 90, or 120 mg) to receive a single dose of KMY tablet or matching placebo under fasting conditions.
  Part B (Multiple Ascending Dose): Participants will be assigned to one of three predefined dose regimens (40 mg QD, 80 mg QD, or 40 mg BID) to receive KMY tablet or matching placebo for 7 consecutive days under fasting conditions.
  Part C (Food Effect): All participants will receive a single dose of 60 mg KMY tablet in a two-period, two-sequence crossover design, once under fasting conditions and once after a high-fat, high-calorie meal.
  This arm includes all participants who receive the active KMY tablet, regardless of the study part, dose level, or fed/fasting condition.
  Interventions: Drug: KMY Tablets
- KMY Tablets Placebo (Placebo Comparator): Participants will receive a placebo tablet identical in appearance to the KMY tablet but containing no active ingredient. The placebo is used only in the randomized, double-blind, controlled portions of the study (Part A and Part B). Within each dose cohort of Part A and Part B, a subset of participants will be randomized to this arm.
  This arm does NOT include participants from the open-label Part C study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KMY Tablets — KMY Tablets is an investigational drug product. This study evaluates its safety, tolerability, and pharmacokinetics in healthy subjects.
  Other Names: Investigational Product
  Arms: KMY Tablets
Drug: Placebo — A placebo tablet matching the appearance of the active KMY Tablets. It contains no active pharmaceutical ingredient.
  Other Names: Placebo matching KMY Tablets
  Arms: KMY Tablets Placebo

SUMMARY:
This is a Phase Ia, randomized, double-blind, placebo-controlled study conducted in healthy subjects. The study plans to enroll a total of 120 participants, with both males and females included in all parts.

The trial consists of three distinct parts:

Part A (Single-Ascending Dose, SAD): A total of 72 subjects will be enrolled to evaluate the safety, tolerability, and pharmacokinetics of single oral doses of KMY Tablets.

Part B (Multiple-Ascending Dose, MAD): A total of 36 subjects will be enrolled to evaluate the safety, tolerability, and pharmacokinetics of multiple oral doses of KMY Tablets.

Part C (Food-Effect): A total of 12 subjects will be enrolled to assess the impact of a high-fat, high-calorie meal on the pharmacokinetic profile of KMY Tablets.

The primary objectives are to evaluate the safety and tolerability of single and multiple doses of KMY Tablets and to assess the food effect on its pharmacokinetics. The secondary objectives include characterizing the single- and multiple-dose pharmacokinetics, investigating the drug's metabolism and excretion, and evaluating the safety and tolerability in the fed state. Exploratory pharmacodynamic parameters may also be investigated.

DETAILED DESCRIPTION:
This is a single-center, Phase Ia, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, and pharmacokinetics of KMY Tablets in healthy subjects. The study consists of three parts: a Single-Ascending Dose part, a Multiple-Ascending Dose part, and a Food-Effect part. A total of 120 subjects will be enrolled. The primary objectives are to assess the safety and tolerability profile and to investigate the effect of food on pharmacokinetics. Secondary objectives include characterizing the single- and multiple-dose pharmacokinetic profiles and investigating the metabolism and excretion of KMY Tablets

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female participants aged 18 to 45 years (inclusive).
2. Male participants weigh ≥50.0 kg; female participants weigh ≥45.0 kg. Body Mass Index (BMI) is between 19.0 and 26.0 kg/m² (inclusive).
3. Participants agree to use effective contraception from screening until a specified period after the last dose and have no plan for pregnancy, sperm donation, or egg donation.
4. Voluntarily participate in the trial, fully understand the study, sign the informed consent form, and are able to comply with the study procedures.

Exclusion Criteria：

1. Known history of allergy to the active ingredient, excipients of the investigational drug, or related compounds; or allergic constitution (e.g., allergy to two or more drugs or foods).
2. History or presence of severe chronic diseases of the cardiovascular, hepatic, renal, respiratory, hematological, endocrine, immune, psychiatric, or neurological systems within the past year, which in the investigator's judgment may compromise participant safety or study integrity.
3. Abnormal and clinically significant findings in vital signs, physical examination, laboratory tests (hematology, blood chemistry, urinalysis, coagulation), or 12-lead ECG at screening, as judged by the investigator.
4. Use of any medications (including prescription, over-the-counter, or herbal medicines) or health supplements within a specified period (e.g., 2 weeks) prior to screening.
5. Participation in another clinical trial (drug or medical device) or use of any other investigational drug within a specified period (e.g., 3 months) prior to screening.
6. History of drug abuse or positive urine drug screen.
7. Donation or loss of ≥400 mL of blood, or receipt of blood products, within a specified period (e.g., 6 months) prior to screening.
8. History of alcohol abuse, inability to abstain from alcohol during the study, or positive alcohol breath test.
9. Smoking more than a specified number of cigarettes per day (e.g., 5) within a specified period prior to screening, or inability to cease use of tobacco products during the study.
10. Intolerance to venipuncture or history of needle or blood phobia.
11. Any other condition that, in the investigator's opinion, may pose a risk to the participant or interfere with the evaluation of study results.

    Additional Exclusion Criteria for Female Participants:
12. Pregnant or lactating women, or women with a positive pregnancy test.
13. Unwilling to use effective contraception during the study and for a specified period thereafter.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-11-07 (Estimated); Study Completion 2026-11-07 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability: Incidence of Treatment-Emergent Adverse Events (TEAEs) | From first dose of study drug up to 7 days after the last dose (assessed up to approximately 4 weeks).
  The number and percentage of participants with all-cause adverse events (AEs), including serious adverse events (SAEs) and AEs leading to study drug discontinuation. Severity will be graded according to NCI CTCAE v5.0.
  (Note: Specify the exact grading scale you use, e.g., NCI CTCAE v5.0)
Food Effect: Maximum Observed Plasma Concentration (Cmax) of KMY Tablets | Pre-dose, and at multiple timepoints up to 72 hours post-dose in each study period (Period 1 and Period 2).
  The maximum observed plasma concentration (Cmax) of KMY Tablets following a single oral dose under fed (high-fat, high-calorie meal) conditions compared to fasting conditions.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve (AUC) of KMY Tablets | Pre-dose, and at multiple timepoints up to 72 hours post-dose.
  The area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC0-t) and extrapolated to infinity (AUC0-∞) following single and multiple doses of KMY Tablets.
Time to Maximum Plasma Concentration (Tmax) of KMY Tablets | Pre-dose, and at multiple timepoints up to 72 hours post-dose.
  The time to reach the maximum observed plasma concentration (Cmax) following single and multiple doses of KMY Tablets.
Cumulative Excretion of KMY and its Metabolites | Urine/feces collection at intervals from 0 to 72 hours post-dose.
  The cumulative amount of KMY and its major metabolites excreted in urine and feces (if collected) over a specified time period.

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Yu, PhD, Principal Investigator — Suzhou Municipal Hospital
Locations (1):
- Suzhou Municipal Hospital, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No